CLINICAL TRIAL: NCT05308836
Title: Phase I Open Label Clinical Trial to Evaluate Safety of Adipose Derived Mesenchymal Stem Cell Transplantation for Type 1 Diabetes Treatment
Brief Title: Evaluate Safety of Adipose Derived Mesenchymal Stem Cell Transplantation for Type 1 Diabetes Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Collaborators: Gwoxi Stem cell applied technology Company (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISC20.01
Record Dates: First submitted 2022-02-25; First posted 2022-04-04 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes Adipose-derived mesenchymal stem cell
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adipose-derived messenchymal stem cell (AD-MSC) (Experimental): Intervention: Intravenousling (IV) AD-MSC in 10 patients with type 1 diabetes mellitus.
  Interventions: Combination Product: adipose-derived messenchymal stem cell

INTERVENTIONS:
Combination Product: adipose-derived messenchymal stem cell — Collaborative research program between Vinmec Research Institute of Stem Cell and Gene Technology with the National Yang-Ming University in Taiwan The adipose mesenchymal stem cell line (GXIPC1) was collected from healthy donors who have screened for infectious diseases and then multiplied in large numbers. These products were produced following the GMP laboratory system and approved by Taiwan FDA for preclinical and clinical trials with completed certificates

SUMMARY:
The purpose of this study is to evaluate the safety of intravenously (IV) administered adipose-derived mesenchymal stem cell (AD-MSC) in patients with type 1 diabetes mellitus (T1D)

DETAILED DESCRIPTION:
Adipose derived mesenchymal stem cells (AD-MSCs) has many advantages, i.e. the greater ease of access and harvesting by means such as subcutaneous lipoaspiration, a much less painful procedure than harvesting bone marrow stem cells, and a much less ethical concern because they are harvested from autologous fat. The purpose of this study is to evaluate the safety of intravenously (IV) administered adipose-derived mesenchymal stem cell (AD-MSC) in treatment 10 patients with type 1 diabetes mellitus (T1D) at Vinmec International Hospital, Hanoi, Vietnam.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed T1D (according to the instructions of the Ministry of Health No: 5481/QD-BYT dated December 30, 2020)
* Aged from 5 years and over.
* The time from the diagnosis of type 1 diabetes to enrollment ≤ 12 months.
* Blood testing conducted at the time of diagnosis:

  * Fasting blood glucose ≥ 7 mmol / L,
  * HbA1C ≥ 6.5%.
  * Have at least one antibodies associated with T1D such as ICA; GAD; ZnT8 or IAA.
* At the time of screening at Vinmec for study enrollment, patients are actively managing their blood glucose levels with insulin.
* The patient does not have other serious acute illness requiring treatment
* The patient agrees to use stem cell transplant for treatment
* The patient's parent (parent or legal guardian) can read, write, understand the ICF form and agree to sign a consent to participate in the study.

Exclusion Criteria:

* Having evidence related to renal dysfunction: creatinine > 1.5 mg/dl or (>133 mmol/L) for boys, creatinine > 1.4 mg/dl or (>124 mmol/L) for girls
* In case of kidney failure. Proteinuria within the range of nephrotic syndrome (>3.5 g/day or ratio of protein/creatinine in urine >2.7)
* In case of kidney failure
* Having severe infection or infected with hepatitis B virus, hepatitis C virus, HIV virus, or tuberculosis
* Cardiovascular disease, respiratory disease (pulmonary, fibrosis, chronic respiratory failure), liver disease, cancer or neurological disease
* Blood clotting disorders (INR> 1,5, PTT> 40, PT> 15).
* Taking any anticoagulant
* Taking systemic steroids
* Participate in another clinical study involving experimenting drugs and/or medical equipment
* History of allergic reaction to anesthetic agents and/or antibiotics

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Safety measure | up to the 6-month period following treatment
  Safety is recognized as number of adverse events (AE) and serious adverse events (SAE) appear from the time that patients sign in ICF

SECONDARY OUTCOMES:
HbA1c | up to the 6-month period following treatment
  A hemoglobin A1c (HbA1c) test measures the amount of blood sugar (glucose) attached to hemoglobin
Fasting blood glucose (FPG) | up to the 6-month period following treatment
  Fasting blood glucose (FPG) measures the levels of glucose (sugar) in the blood
C-peptide levels | up to the 6-month period following treatment
  C-peptide levels
Blood insulin | up to the 6-month period following treatment
  Blood insulin
Insulin dose | up to the 6-month period following treatment
  Insulin dose

CONTACTS AND LOCATIONS:
Overall Officials: Liem T Nguyen, Prof, Principal Investigator — Vinmec Research Institute of Stem Cell and Gene Technology
Locations (1):
- Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Y, Chen W, Feng B, Cao H. The Clinical Efficacy and Safety of Stem Cell Therapy for Diabetes Mellitus: A Systematic Review and Meta-Analysis. Aging Dis. 2020 Feb 1;11(1):141-153. doi: 10.14336/AD.2019.0421. eCollection 2020 Feb. PMID 32010488
- [Background] Araujo DB, Dantas JR, Silva KR, Souto DL, Pereira MFC, Moreira JP, Luiz RR, Claudio-Da-Silva CS, Gabbay MAL, Dib SA, Couri CEB, Maiolino A, Rebelatto CLK, Daga DR, Senegaglia AC, Brofman PRS, Baptista LS, Oliveira JEP, Zajdenverg L, Rodacki M. Allogenic Adipose Tissue-Derived Stromal/Stem Cells and Vitamin D Supplementation in Patients With Recent-Onset Type 1 Diabetes Mellitus: A 3-Month Follow-Up Pilot Study. Front Immunol. 2020 Jun 2;11:993. doi: 10.3389/fimmu.2020.00993. eCollection 2020. PMID 32582156